CLINICAL TRIAL: NCT02704884
Title: Microbial Soy Milk Consumption, Inflammation and Renal Function Among Type 2 Diabetic Patients With Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Makan Pourmasoumi, MSc student, Principal Investigator, Department of Community Nutrition, School of Nutrition and Food Science, Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 394733
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Type II Diabetic Patients With Nephropathy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- probiotic soy milk (Experimental): consume a diet containing 200 ml/day probiotic soy milk in intervention group
  Interventions: Dietary Supplement: probiotic soy milk
- soy milk (Active Comparator): 200 ml/day soy milk in the control condition
  Interventions: Dietary Supplement: probiotic soy milk

INTERVENTIONS:
Dietary Supplement: probiotic soy milk

SUMMARY:
The aim of the present study was to determine the effects of fortified soy milk with L. planetarium A7 on a cytokine receptor, an adipokine and renal function biomarkers in type II diabetic patients with nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Type 2 diabetic patients with stages 1 and 2 of nephropathy (defined as meeting criteria including fasting blood glucose >126 mg/dL, hypoglycemic agents, or insulin intake, proteinuria >300 mg/day, and glomerular filtration rate >90 mL/min)

Exclusion Criteria:

* pregnancy or lactating in women
* allergy or intolerance to soy milk or avoidance of soy milk consumption
* smoking, alcoholism
* recent antibiotic therapy and using of supplements containing vitamins and minerals
* any medical condition such as inflammatory bowel disease, infection, liver disease and rheumatoid arthritis.

Ages: 32 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
inflammatory adipokine- Progranulin (PGRN) | 8 week
  PGRN will determine by commercial sandwich enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's protocols. (Human ELISA kits, Shanghai Crystal Day Biotech Company, China).
cytokine receptor -soluble tumor necrosis factor receptor 1 (sTNFR1), | 8 week
  sTNFR1 will determine by commercial sandwich enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's protocols. (Human ELISA kits, Shanghai Crystal Day Biotech Company, China).
serum levels of Neutrophil gelatinase-associated lipocalin (NGAL) | 8 week
  NGAL will determine by commercial sandwich enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's protocols. (Human ELISA kits, Shanghai Crystal Day Biotech Company, China).
cystatin C (Cys- C) | 8 week
  Cys- C will determine by commercial sandwich enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's protocols. (Human ELISA kits, Shanghai Crystal Day Biotech Company, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Makan Pourmasoumi, Tehran, Iran

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Miraghajani M, Zaghian N, Mirlohi M, Feizi A, Ghiasvand R. The Impact of Probiotic Soy Milk Consumption on Oxidative Stress Among Type 2 Diabetic Kidney Disease Patients: A Randomized Controlled Clinical Trial. J Ren Nutr. 2017 Sep;27(5):317-324. doi: 10.1053/j.jrn.2017.04.004. Epub 2017 May 31. PMID 28579313